CLINICAL TRIAL: NCT06719206
Title: Reduce Sedentary Behavior During Cancer Treatment - the RedSedCan Study
Acronym: RedSedCan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Collaborators: Region Västmanland (Other); Uppsala University (Other); Centrallasarettet Västerås (Other); Uppsala University Hospital (Other); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/1120
Record Dates: First submitted 2024-11-19; First posted 2024-12-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Colorectal Cancer (CRC); Prostate Cancer; Neoadjuvant Therapy; Adjuvant Therapy
Keywords: sedentary behavior; behavior change; intervention; Randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive a digital support intervention
  Interventions: Behavioral: Digital self-management program
- Control (No Intervention): Control condition. Individuals receive the care as usual provided by the healthcare only.

INTERVENTIONS:
Behavioral: Digital self-management program — The program consists of commercially available technologies, e.g. applications including behavour change techniques for reducing sedentary behavior (SB) (i.e. self-monitorization of physical activity, reminders for breaking SB/doing physical activity, and providing feedback on physical activity/breaks from SB) and a webpage containing information and tips (provided in short videos and text) regarding how to reduce SB. The participants will be receive help with setting goals for reducing time spent in sedentary/being active and help with planning for what activities to do to replace time in sedentary. Participants will then have access to the webpage and download the application to their smartphones. Follow-up meetings with the physiotherapist (digital or physical) will be conducted after 2, 8 and 12 weeks after start of intervention.
  Arms: Intervention

SUMMARY:
Summary

Reducing sedentary behavior during treatment is important to reduce the risk of future health problems in individuals undergoing cancer treatment. Therefore, the goal of this project is with a multicenter randomised controlled design investigate whether a digital support intervention during ongoing neo- or adjuvant cancer treatment for breast, prostate or colon cancer is effective in reducing sedentary lifestyle and improving well-being in the short and long term.

DETAILED DESCRIPTION:
Description of the project

This project is about investigating the effect of a digital support intervention to reduce sedentary behavior in people with breast, prostate, or colorectal cancer during neo- or adjuvant cancer treatment. The digital support intervention has been developed with patients and researchers and consists of existing high-quality technology that provides support for setting and following goals. The people who use the digital support intervention also receive support from a physiotherapist to set goals for reduced sedentary time and get to choose which activities will replace the time spent sedentary.

The goal of the project

The goal of the project is to investigate the effects of a digital support intervention on reduced sedentary and well-being during ongoing cancer treatment, both in the short and long term. In addition, the project will study the health-economic effects, and climate benefits of using the digital support intervention. By focusing on reducing a sedentary lifestyle and replacing it with daily activities and/or physical activity, the health of individuals is expected to be positively affected in the short term through, for example, increased well-being and reduced side effects from cancer treatment, and the long term through a reduced risk of developing complications and new illness related to the cancer treatment, such as cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with breast, prostate, or colorectal cancer planned for or resently started neo- or adjuvant treatment (e.g. chemotherapy, radiotherapy, endocrine treatment) at the hospitals in Uppsala and Västerås, Sweden.

Exclusion Criteria:

* Individuals diagnosed with dementia.
* Individuals diagnosed with severe psychiatric disease.
* Individuals with severe loss of vision, or communicative ability.
* Individuals who cannot walk independently indoors with or without a walking aid.
* Individuals completed treatment for other cancer diseases less than 12 months ago or not recovered from previous cancer treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Sedentary behavior time | At baseline, 3-months, 6 months, 12 months and 24 months. Axivity is worn for 7 consecutive days at each measurement point.
  The Axivity accelerometer is used for measuring the primary outcome of sedentary time, i.e. mean time spent in sedentary behavior/day.

SECONDARY OUTCOMES:
Sedentary behavior bouts | At baseline, 3-months, 6 months, 12 months and 24 months. Axivity is worn for 7 consecutive days at each measurement point.
  The Axivity accelerometer is used for measuring sedentary bouts, i.e. mean number of bouts/day and mean bouts time/day.
Physical activity | At baseline, 3-months, 6 months, 12 months and 24 months. Axivity is worn for 7 consecutive days at each measurement point.
  The Axivity accelerometer is used for measuring physical activity mean time/day and mean time spent in low-, moderate and high intensity physical activity.
Health-related quality of life | At baseline, 3-months, 6 months, 12 months and 24 months.
  Patient reported health related quality of life will be assessed with European Organization for Research and Treatment of Cancer QLQ C 30 and diagnose specific modules BR23, PR26 and CR29.
Health-related quality of life | At baseline, 3-months, 6 months, 12 months and 24 months.
  Patient reported health related quality of life will be assessed with EQ5D, and used for calculation of Quality Adjusted Life Years.
Cancer related fatigue | At baseline, 3-months, 6 months, 12 months and 24 months.
  Patient reported outcome cancer related fatigue is measured with Brief Fatigue Inventory.
Fear of movement | At baseline, 3-months, 6 months, 12 months and 24 months.
  Patient reported outcome Fear of movement is assessed with Cancer specific Tampa Scale for Kinesiophobia.
Changes in health | At 3-months, 6 months, 12 months and 24 months.
  Patient reported outcome Changes in health is assessed with Patient Global Impression of Change Scale.
Work ability | At baseline, 3-months, 6 months, 12 months and 24 months.
  Selected and adapted questions from Work Ability Index are used for assessing patient reported outcome work ability.
Self-efficacy for reducing sedentary behavior | At baseline, 3-months, 6 months, 12 months and 24 months.
  Study specific question is used for assessing patient reported outcome of Self-efficacy for reducing sedentary behavior.
Perceived support from peers | At baseline, 3-months, 6 months, 12 months and 24 months.
  Study specific question is used for assessing patient reported outcome of Perceived support from peers.

OTHER OUTCOMES:
Demographic variables | Baseline
  Study specific questions
Diagnoses | At baseline
  Data regarding cancer diagnose and if any, co-morbid conditions, are gathered from medical records or Swedish national quality registers.
Cancer treatment | At baseline, 3-months, 6 months, 12 months and 24 months.
  Data regarding planned and received oncological and surgical cancer treatment (type, dose, treatment start and end date of treatment) and any treatment related side-effects are gathered from medical records and Swedish quality registers.
Health care costs | At baseline, 3-months, 6 months, 12 months and 24 months.
  Data regarding outpatient visits, hospitalization and prescribed medication is gathered from Swedish national quality registers.
Costs of intervention | At baseline, 3-months, 6 months, 12 months and 24 months.
  Data regarding cost of application use and any cost for physical activity is gathered from study records and patient reported by study specific questions.
Sick leave | At baseline, 3-months, 6 months, 12 months and 24 months.
  Data regarding sick leave, i.e. total number of days being on sick leave gathered from the Swedish insurance fund (data on sick leave more than 14 days) and patient reported study specific questions (data on sick leave less than 14 days). Data will be gathered from 6 months prior baseline (study specific questions are administered at baseline and register data will be gathered at baseline but will include any data 6 months prior baseline).
Adherence | At baseline, 3-months, 6 months, 12 months and 24 months.
  Adherence to the intervention is assessed by Axivity accelometer and patient reported study specific questions.
Green house gas emissions | At baseline, 3-months, 6 months, 12 months and 24 months.
  Green house emissions will be compared between the intervention and control group and estimated using a life cycle analysis of the technology used in the intervention, self-reported changes in climate behavior, and emissions from healthcare.

CONTACTS AND LOCATIONS:
Overall Officials: Petra von Heideken Wågert, Professor, Principal Investigator — Mälardalen University
Locations (2):
- Sweden (2):
  - Akademiska sjukhuset, Uppsala
  - Västmanlands sjukhus, Västerås

IPD SHARING:
Plan to Share IPD: No
Individual medical information may not be shared with other researchers if the research questions are not within the scope of the current approved Swedish Ethical Review Board application (and any amendments) for this research. Only pseudonymous information may be shared after approval has been provided from the Swedish Ethical Review Board.

REFERENCES:
- See also: Offical study web page at Mälardalens University — https://www.mdu.se/en/malardalen-university/research/research-projects/reduce-sedentary-behavior-during-cancer-treatment---the-redsedcan-study